CLINICAL TRIAL: NCT05357339
Title: The Effect of Fluid Resuscitation with 20% Albumin Versus Crystalloid on the Microcirculation of Patients with Sepsis
Brief Title: Microcirculation Properties of Albumin for Fluid Resuscitation in Septic Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rachael Cusack (Other)
Collaborators: Grifols Biologicals, LLC (Industry)
Responsible Party: Sponsor-Investigator, Rachael Cusack, ICU PhD Candidate, St. James's Hospital, Ireland
Organization: St. James's Hospital, Ireland (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MICALB21
Record Dates: First submitted 2022-01-19; First posted 2022-05-02 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Sepsis, Severe; Sepsis; Septic Shock
Keywords: microcirculation; sidestream dark field
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Albumins; Crystalloid Solutions

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional 20% Albumin (Experimental): Septic patients requiring a fluid bolus randomised to receive 100ml 20% albumin as boluses until they are stable or no longer require fluid resuscitation.
  Interventions: Other: 20% Albumin
- Control Crystalloid (Active Comparator): Septic patients requiring a fluid bolus randomised to receive 250ml boluses of crystalloid fluid until they no longer require fluid resuscitation.
  Interventions: Other: Crystalloid

INTERVENTIONS:
Other: 20% Albumin — 100ml boluses 20% Albumin
  Arms: Interventional 20% Albumin
Other: Crystalloid — 100ml bolus of crystalloid
  Arms: Control Crystalloid

SUMMARY:
The sublingual microcirculation is impaired in sepsis and septic shock. Sidestream dark field imaging technology has been developed into a clinical tool to help the clinician assess the microcirculation at the bedside. The ideal resuscitation fluid has not been identified. The investigators aim to use this new bedside technology to establish the microcirculation properties of two popular resuscitation fluids.

DETAILED DESCRIPTION:
Sepsis and septic shock are diseases of the microcirculation. Recent developments in microcirculation imaging have illustrated the extent of the impairment of the microcirculation in these diseases of critical care. Heterogenous flow, stagnation and microthrombi can all be seen clearly in the sublingual region using a sidestream dark field imaging device.

One of the key treatments for sepsis and septic shock is timely administration of intravenous fluids. Which fluid is administered is a matter for debate which has not been settled by several large trials. De-resuscitation has become increasingly important as physicians realise the implications and associated risks of excess fluid administration in ICU. Avoiding excess fluid administration at the resuscitation stage is therefore desirable. One of the prevailing theories about the function of albumin or colloid resuscitation is that it remains in the the intravascular space for a longer period of time, thereby continuing to benefit the patient and avoiding administration of excess fluid. However, recently albumin was tested against crystalloid for resuscitation and was shown to be effective but with no improvement in survival.

It is possible, however, that albumin is having an initial beneficial effect at a microcirculation level. Macrohaemodynamic improvements are not necessarily matched by improvements in blood flow and oxygen delivery to cells, this has been referred to as haemodynamic incoherence.

This randomised, prospective study aims to compare crystalloid and albumin resuscitation at a microcirculation level.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis; suspected source of infection, tachycardia, tachypneic, hyperlactatemia, hypotensive requiring vasopressors, febrile >38.5degrees Celsius
* Fluid responsive; pulse pressure variability >10% or passive leg raise positive

Exclusion Criteria:

* Fluid overloaded; pulmonary oedema, significant peripheral oedema
* Heart Failure, cardiogenic shock, recent MI
* Receiving regular albumin 20%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Microcirculation parameters in response to a fluid bolus | Baseline at recruitment before fluid given, during bolus, after bolus: immediately after, 60 minutes after and 24 hours after to determine if immediate, delayed or sustained change in microcirculation parameters is influenced by fluid bolus
  functional capillary density, perfused capillary density after fluid bolus Proportion Perfused vessels Microvascular Flow Index Total Vessel Density

SECONDARY OUTCOMES:
Duration of vasopressor administration | 28 days
Duration of Mechanical ventilation | 28 days
ICU length of stay | though to stud completion; up to 1 year
28 day mortality | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- St James's Hospital, Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cusack R, Rodriguez A, Cantan B, Miskolci O, Connolly E, Zilahi G, Coakley JD, Martin-Loeches I. Albumin Enhances Microvascular Reactivity in Sepsis: Insights from Near-Infrared Spectroscopy and Vascular Occlusion Testing. J Clin Med. 2025 Jul 14;14(14):4982. doi: 10.3390/jcm14144982. PMID 40725675
- [Derived] Cusack RAF, Rodriguez A, Cantan B, Garduno A, Connolly E, Zilahi G, Coakley JD, Martin-Loeches I. Microcirculation properties of 20 % albumin in sepsis; a randomised controlled trial. J Crit Care. 2025 Jun;87:155039. doi: 10.1016/j.jcrc.2025.155039. Epub 2025 Feb 27. PMID 40020556